CLINICAL TRIAL: NCT03955692
Title: The Efficacy of Cathodal Transcranial Direct Current Stimulation in Children and Adolescents With Attention-deficit Hyperactivity Disorder
Brief Title: The Efficacy of Cathodal tDCS in ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MU-IRB 2017/046.2002
Record Dates: First submitted 2017-11-16; First posted 2019-05-20 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Cathodal tDCS will be applied over the left DLPFC (F3) according to the 10-20 EEG electrode systems and the anode will be placed over the right supraorbital (Fp2), using rectangular saline-soaked sponge pads 35 cm2. The current intensity of 1.5 mA will be used for 15 mins for a session.
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): Cathodal tDCS will be applied over the left DLPFC (F3) according to the 10-20 EEG electrode systems and the anode will be placed over the right supraorbital (Fp2), using rectangular saline-soaked sponge pads 35 cm2. The current intensity of 1.5 mA will flow continuously only 120 seconds. The electrode will be attached until the end of stimulation even the current flows only at the beginning.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Five sessions (active/sham) will be held on five consecutive days. The parameter of electrode size, current strength and current duration were previously tested for safety in children

SUMMARY:
The purpose of this study is to investigate the effectiveness of five sessions of cathodal tDCS over the left DLPFC on inhibitory control/response inhibition in children and adolescents with ADHD. Investigators hypothesize that multiple sessions of cathodal tDCS will induce a greater and long-term effect on inhibitory response in children and adolescents with ADHD.

DETAILED DESCRIPTION:
Attention-deficit hyperactivity disorder (ADHD) is one of neural development disorder that characterized by a persistent pattern of inattention, impulsivity and hyperactivity. This disorder begins in childhood and often lasts into adulthood. Rates of ADHD diagnosis have been rising in recent years, a prevalence estimates from 3-7% of childhood worldwide. A recent national prevalence shows that 8.1% of Thai primary school-age children are affected by ADHD . Pharmacological treatment used in ADHD is well-established, however, each patient responds to medication differently and treatment in some of them are limited by side effect and abuse of medication.

In the last decade, transcranial direct current stimulation (tDCS) has received a surge of interest in clinical research since it could modulate cortical excitability and induce plasticity in human brain. The device sends a constant low direct current (e.g. 1-2 mA) delivered to the area of interest through the electrodes. This induces shifts in neuronal resting membrane potential changing cortical excitability. Based on the polarity-specific effects, anodal tDCS increases cortical excitability and cathodal tDCS decreases cortical excitability. To change the cortical excitability, tDCS differs from other brain stimulation techniques such as transcranial magnetic stimulation (TMS) in that it does not cause action potentials in cortical neurons, but rather induces shifts in neuronal resting membrane potential. This is considered to induce a lesser or no risk of a seizure. Given its advantages such as painlessness, safety, easiness to use, and low-cost, a number of tDCS studies has been increasing in the last decade particularly in motor rehabilitation and neuropsychiatric disorders such as depression, autism and schizophrenia with a positive and safety reports in adult and pediatric populations. Possible after-effect of tDCS has been also reported in motor and psychological disorders that opens a way to use tDCS as a therapeutic tool.

The most accepted theory of neural basis of ADHD is deficient of inhibitory control resulting in executive dysfunction. Inhibitory control or response inhibition is key feature of self-control and can be defined as ability to inhibit prepotent actions. Several evidences reveal a physiological association between the prefrontal cortex and its subcortical connection with the pathophysiology of ADHD. Neuroimaging studies demonstrate that regions of the right dorso-lateral prefrontal cortex (DLPFC) play a role in the inhibition of motor response. During preforming an inhibitory task that is usually used to evaluate the efficiency of response inhibition such as stop-signal and go/no-go tasks, this area become active in healthy individual, while in ADHD showed hypo-activation compared to control.

Evidences showed that the task performance in stop-signal and go/no-go tasks can be influenced by tDCS application to the DLPFC in healthy subjects. It was recently reported that a single session of cathodal tDCS, using a single session of 1.5 mA for 15 minutes over the left DLPFC improved their ability to inhibit themselves by do not response to no-go stimulus during go/no-go tasks compared to anodal and sham conditions in adolescents with ADHD. It was postulated that the inter-hemispheric inhibition (IHI) between two regions (left and right DLPFC) might play a role in this finding. Based on the possibility that cathodal stimulation decreases excitability and thus IHI drive from the left DLPFC is decreased, facilitating activity of the right DLPFC where is involved in inhibition of motor response as demonstrated by neuroimaging studies. Using a single session of oscillatory tDCS during early sleep, memory consolidation and reaction times in a go/no-go task were improved on the next day in children with ADHD. This is an argument to explore its possible therapeutic effect in long-term use. Five tDCS sessions for five consecutive days was reported to be safe and improves aspect of attention in children and adolescents with ADHD, however, its after-effect in this population is unknown. In patients with depressive disorder, multiple sessions of tDCS over the left DLPFC for five or ten days has been demonstrated to decrease depressive symptoms and lasted for a month. It was reported in patient with depressive disorder that after five days of tDCS sessions on alternative day did not show an improvement, positive results was observed after 10 days. This suggests that a longer observation period is probably required to detect a true tDCS effect.

The use of electrophysiological techniques, especially of event-related potentials (ERP) measured by means of electroencephalography (EEG) allows for analysis of neural change accompanying inhibitory process in the brain. Two ERP components, the no-go N2 and P3 that are the most commonly studied in go/no-go tasks have been linked to response conflict and response inhibition. Studies have reported lower N2 and P3 amplitudes during go/no-go tasks in children and adolescents with ADHD.

To expand current information on tDCS as an emerging treatment for ADHD patients, in this study, investigators will investigate the effectiveness of multiple sessions of cathodal tDCS over the left DLPFC on inhibitory control in children and adolescents with ADHD. tDCS (cathodal/sham) will be applied every day for five consecutive days. Behavioral and neurophysiological parameters using an inhibitory task (go/no-go tasks) and the no-go N2 and P3 ERP components will be measured before tDCS, immediately after 5 sessions of tDCS, one week later, and one month after treatment onset.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents aged 7 to 16 years with suspected ADHD according to the Diagnostic and Statistical Manual of Mental Disorders-5th edition (DSM-5TM). Diagnostic confirmation will be performed by pediatric neurologist or psychologist.
2. Right-handed
3. Free of any neurological antecedent, unstable medical conditions such as epilepsy; although tDCS is believed to induce very less or no risk of seizure and epileptic seizure have never been reported in tDCS study even in a study with active epilepsy.

Exclusion Criteria:

1. Be unable to understand the instruction
2. No clear neurological antecedent history
3. Presence of intracranial metal implantation, cochlea implant, or cardiac pacemaker
4. Motor or perceptual handicap that would prevent using the computer program
5. For patients who under medication, poor-adjusted to their medication, type and dosage of medication is changed less than 4 weeks prior to the start
6. Subjects are participating in the other protocol or receiving alternative treatment such transcranial magnetic stimulation.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change of accuracy rate | Change from baseline to Day 0 after tDCS (T1)
  Accuracy rate from go/no-go tasks
Change of accuracy rate | Change from Day 0 to 1 week after tDCS (T2)
  Accuracy rate from go/no-go tasks
Change of accuracy rate | Change form 1 week to 1 month after tDCS (T3)
  Accuracy rate from go/no-go tasks
Change in the amplitude of ERP recording | Change from baseline to Day 0 after tDCS (T1)
  The amplitude of the ERP components (N2 and P3) in average will be use as outcome measures to evaluate response inhibition.
Change in the amplitude of ERP recording | Change from Day 0 to 1 week after tDCS (T2)
  The amplitude of the ERP components (N2 and P3) in average will be use as outcome measures to evaluate response inhibition.
Change in the amplitude of ERP recording | Change form 1 week to 1 month after tDCS (T3)
  The amplitude of the ERP components (N2 and P3) in average will be use as outcome measures to evaluate response inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Wanalee Klomjai, PhD, Principal Investigator — Mahidol University
Locations (1):
- Faculty ofPhysical Therapy, Mahidol University, Salaya, Nakonpathom, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klomjai W, Siripornpanich V, Aneksan B, Vimolratana O, Permpoonputtana K, Tretriluxana J, Thichanpiang P. Effects of cathodal transcranial direct current stimulation on inhibitory and attention control in children and adolescents with attention-deficit hyperactivity disorder: A pilot randomized sham-controlled crossover study. J Psychiatr Res. 2022 Jun;150:130-141. doi: 10.1016/j.jpsychires.2022.02.032. Epub 2022 Mar 2. PMID 35367657